CLINICAL TRIAL: NCT07292883
Title: Accelerated Deep Transcranial Magnetic Stimulation for Smoking Cessation
Brief Title: Accelerated dTMS Smoking Cessation
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Waypoint Centre for Mental Health Care (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5240
Record Dates: First submitted 2025-11-20; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Tobacco Use Disorder; Addiction Nicotine
Keywords: addiction; smoking cessation; Transcranial Magnetic Stimulation; Accelerated Repetitive Transcranial Magnetic Stimulation
MeSH Terms: conditions — Tobacco Use Disorder; Behavior, Addictive; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Accelerated Repetitive Transcranial Magnetic Stimulation (Experimental): Bilateral Accelerated Repetitive Transcranial Magnetic Stimulation targeting the insula and prefrontal cortex using H4 coil
  Interventions: Device: Bilateral deep accelerated repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: Bilateral deep accelerated repetitive transcranial magnetic stimulation — Accelerated Repetitive Transcranial Magnetic Stimulation (aTMS) is a type of treatment that will be used to target the bilateral insular cortex and prefrontal cortex using the Health Canada-approved H4 coil. The purpose is to test its feasibility on smoking abstinence. While convention rTMS methods involves one session daily over several weeks, aTMS delivers multiple sessions per day. Using the H4 deep aTMS, this study will implement 20 sessions over five consecutive days (four sessions daily).
  Other Names: Deep TMS; Accelerated TMS; Repetitive TMS

SUMMARY:
The goal of this clinical trial is to examine whether a 5-day course of bilateral accelerated deep transcranial magnetic stimulation (aTMS) is a feasible treatment to help adults (18-65) with Tobacco Use Disorder to quit smoking. This study aims to enroll 30-40 participants and will examine treatment tolerability, treatment acceptability, participant retention, and adherence to scheduled treatment sessions.

There are two key objectives and hypotheses:

Objective 1: To evaluate whether a 1-week course of bilateral aTMS (4 sessions per day for 5 days) is feasible and tolerable as a smoking cessation treatment.

Hypothesis 1: Feasibility will be demonstrated by acceptable tolerability, acceptability, retention, and adherence, with a practical target of 30 out of 40 participants completing the treatment.

Objective 2: To explore how aTMS affects smoking outcomes, including:

* Point-prevalence abstinence at end of treatment and at Weeks 3, 5, and 9.
* Prolonged/continuous abstinence at Weeks 13 and 26.
* Craving, cigarettes per day, and dependence severity. Hypothesis 2: Participants will show improvements on these outcomes from post-treatment through follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older;
2. Tobacco use disorder as assessed by DSM-5;
3. Fagerstrom Test of Nicotine Dependence (FTND) ≥ 4;
4. Reported motivation to quit within 30 days as assessed using the Contemplation Ladder score of ≥ 7;
5. Must sign and date the informed consent form;
6. Stated willingness to comply with all study procedures.
7. Able to communicate in English.

Exclusion Criteria:

1. Reported smoking abstinence in the 3 months preceding screening visit;
2. Current use of other smoking cessation aids;
3. Contraindication to rTMS;
4. Pregnancy, trying to become pregnant or breastfeeding;
5. Current or recent history of cerebrovascular disease;
6. Unstable major psychiatric disorder(s) (i.e. Axis I Disorders) that would prevent participation in the study at PI (or its delegate) discretion;
7. Serious current or personal history of medical condition/disease (neurological disorders, brain lesions, multiple sclerosis, head trauma, loss of consciousness, hearing loss, etc.) preventing same inclusion as per PI (or its delegate) discretion;
8. Current, personal history or family history of seizures;
9. Concomitant use of medication that lowers seizure threshold, such as clozapine;
10. Concomitant use of more than 2 mg lorazepam (or an equivalent) or any anticonvulsants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Who Discontinue Accelerated dTMS Due to Side Effects | From week 1 day 1, to week 1 day 5 of treatment week.
  Tolerability will be assessed by calculating the percentage of participants who discontinue the 5-day accelerated dTMS treatment course due to side effects.
TMS Experience Questionnaire Acceptability Scores (Units on a Scale) | From week 1 day 1, to week 1 day 5 of treatment week.
  Acceptability will be assessed using scores on the TMS Experience Questionnaire.
Percentage of Participants Completing the 5-day Accelerated dTMS Treatment Course | From week 1 day 1, to week 5 day 5 of treatment week.
  Retention will be measured by the percentage of enrolled participants who complete the full 5-day accelerated dTMS treatment protocol (4 sessions per day for 5 days). The aim is 30 out of 40 participants (75%) completing the course.
Percentage of Treatment Sessions Attended | From week 1 day 1, to week 1 day 5 of treatment week.
  Adherence will be measured by calculating the percentages of planned accelerated dTMS treatment sessions attended (20 sessions total over 5 days). For each participant, adherence will be calculated as number of sessions attended divided by 20, and then calculating a mean percentage.

SECONDARY OUTCOMES:
The percentage of participants achieving continuous short-term abstinence at follow up | From week 1 day 5 of treatment to week 26.
  Measuring the percentage of participants who achieved 7-day point prevalence abstinence at the end of treatment, week 3, week 5, week 9, week, 13, week 26.
The percentage of participants achieving continuous long-term abstinence at follow up | From week 1 day 1 of treatment to week 26.
  Calculating the percentage of participants who achieved prolonged and continuous absence at week 13 (3 months) and week 26 (6 months).
Change in Tobacco Craving Questionnaire-Short Form (TCQ-SF) Total Score (Units on a Scale) | From baseline to week 26.
  This outcome will examine changes in self-reported cravings using the TCQ-SF. TCQ-SF total scores will be compared from baseline to the end of treatment (week 26) and across follow-up visits (week 3, 5, 9, 13, 26).
Change in Dependence Severity (Units on a Scale) | From baseline to week 26.
  This outcome will examine changes in nicotine dependence severity from baseline to the end of treatment (week 26) and during follow-up visits (week 3, 5, 9, 13) using the Fagerstrom Test for Nicotine Dependence (FTND).
Change in Daily Cigarette Use (Number of Cigarettes per Day) | From baseline to week 26.
  This outcome will examine changes in self-reported cigarette consumption using the Timeline Follow Back method from baseline through follow-ups (week 3, 5, 9, 13) to the end of the study (week 26).

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Le Foll, MD, PhD, MCFP (AM) FCAHS, Principal Investigator — Waypoint Centre for Mental Health Care
Locations (2):
- Canada (2):
  - Waypoint Centre for Mental Health Care, Penetanguishene, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No
There are no plans for use of your study data in other research.

DOCUMENTS (2):
  • Study Protocol (2025-11-05): https://cdn.clinicaltrials.gov/large-docs/83/NCT07292883/Prot_000.pdf
  • Informed Consent Form (2025-05-20): https://cdn.clinicaltrials.gov/large-docs/83/NCT07292883/ICF_001.pdf